CLINICAL TRIAL: NCT03894371
Title: Thermage FLX System to Treat the Face, Neck, and Eyelids for Correction of Mild to Moderate Skin Laxity.
Brief Title: Thermage FLX System to Treat the Face, Neck, and Eyelids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nashville Centre for Laser and Facial Surgery (Other)
Collaborators: Bausch Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-4225
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Facial Skin Laxity

STUDY DESIGN:
Intervention Model Description: Thermage FLX System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thermage (Other): Subjects will undergo treatment with the Thermage FLX system using a 900 pulse, 4cm2 Total Tip to treat the face and neck and a 450 pulse, 0.25cm2 tip to treat the upper and lower eyelids.
  Interventions: Device: Thermage FLX

INTERVENTIONS:
Device: Thermage FLX — Thermage FLX system for the correction of mild to moderate laxity of the skin of the face, neck, and eyelids.

SUMMARY:
25 subjects Fitzpatrick skin type I-VI with mild to moderate laxity of the skin of the face, neck, and eyelids will be enrolled. All subjects will undergo treatment with the Thermage FLX system using a 900 pulse, 4cm2 Total Tip to treat the face and neck and a 450 pulse, 0.25cm2 tip to treat the upper and lower eyelids.

DETAILED DESCRIPTION:
Face/neck: Using a 900 pulse 4.0cm2 Total Tip, 450 pulses will be placed on one half of face/neck on average-large size face, 450 on the other half. Pulses to be placed using several initial passes throughout the treatment zones followed by any remaining pulses to problem areas, as determined by the Investigator. On a petite-small size patient, less pulses may be used on each half of treatment area, at the discretion of the Treating Investigator. Treatment will be performed in the standard manner titrating energy to a subjective discomfort of 2-3 on a 4-point scale, using generous amounts of coupling fluid, and placing return pad on the lower back.

Eyes: Plastic corneoscleral protective lenses will be ised when the eyelids are treated. Using a 450 pulse 0.25cm2 eye tip, 225 pulses will be placed on one eye, 225 on the other eye. Pulses to be placed using several initial passes throughout the treatment zones, followed by any remaining pulses to problem areas, as determined by the Investigator. Treatment will be performed in the standard manner titrating energy to a subjective discomfort of 2-3 on a 4-point scale, using generous amounts of coupling fluid, and placing the return pad on the lower back.

Photographs will be obtained by a professional photographer. Images will be captured at Baseline, and 1, 3, and 6 months post treatment. Treatment outcomes will be assessed at each visit by Subject Global Assessment Improvement Scale (SGAIS), Physician Global Assessment Improvement Scale (PGAIS) abd by blinded assessment of photographs by an independent reviewer. Subjects will be assessed by the Treating Investigator (live) and the non-treating investigator (photographs) using a quartile scale as in the previously published Thermage eyelid trial. Subject satisfaction will also be measured with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 25-70
* Mild to moderate jowling and upper eyelid dermatochalasis
* Willingness to participate in the study
* Understand and complete the informed consent, and willingness to complete all visits. -----Women of childbearing age must have a negative pregnancy test and agree to an acceptable form of birth control for the study duration
* Agreement to use all photographs.

Exclusion Criteria:

* Severe laxity, jowling, and subcutaneous fat
* Severe herniated orbital fat, eyelid ptosis, or other eyelid malposition
* Poor skin quality
* History of neuromodulator use in the previous 6 months
* History of dermal filler use in the past 12 months
* Previous blepharoplasty, rhytidectomy, laser skin resurfacing, trauma or facial reconstructive surgery in the treatment area
* Presence of a beard or facial hair which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessments
* Use of topical facial corticosteroids or prescription retinoids within 1 month of the baseline visit or systemic retinoid treatment within 6 months of the baseline visit
* Presence of any condition, which in the opinion of the Principal Investigator, makes the subject unable to complete the study per protocol or who, in the opinion of the Treating Investigator, should be excluded from the trial.
* History of electronic implanted device, such as, but not limited to, pace maker, internal defibrillator, internal cochlear implant, spinal stimulator, bladder stimulator, etc..
* Currently taking immunosuppressant medications known to interfere with wound healing, response or anti-inflammatory medications (NSAIDS, steroids, other immunosuppressants).
* Patients with underlying diseases that may alter wound healing response (such as diabetes or autoimmune disease).

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Subject Global Aesthetic Improvement Scale | Month 1, post treatment
  The subject will make a direct visual assessment to grade the following indications using the below Quartile Improvement Scale: 0 = No improvement, 1 = Minor/Mild Improvement (0.25%), 2 = Moderate Improvement (26-50%), 3 = Marked Improvement (51-75%), 4 = Very Significant Improvement (76-100%) for Skin Laxity, Skin Texture, and Overall Appearance for the upper face, middle face, lower face, and neck.
Physician Global Aesthetic Improvement Scale | Month 1 post treatment
  The Investigator will make a direct visual assessment to grade the following indications using the below Quartile Improvement Scale: 0 = No improvement, 1 = Minor/Mild Improvement (0.25%), 2 = Moderate Improvement (26-50%), 3 = Marked Improvement (51-75%), 4 = Very Significant Improvement (76-100%) for Skin Laxity, Skin Texture, and Overall Appearance for the upper face, middle face, lower face, and neck.

SECONDARY OUTCOMES:
Subject Global Aesthetic Improvement Scale | Month 3 post treatment
  The subject will make a direct visual assessment to grade the following indications using the below Quartile Improvement Scale: 0 = No improvement, 1 = Minor/Mild Improvement (0.25%), 2 = Moderate Improvement (26-50%), 3 = Marked Improvement (51-75%), 4 = Very Significant Improvement (76-100%) for Skin Laxity, Skin Texture, and Overall Appearance for the upper face, middle face, lower face, and neck.
Physician Global Aesthetic Improvement Scale | Month 3 post treatment
  The Investigator will make a direct visual assessment to grade the following indications using the below Quartile Improvement Scale: 0 = No improvement, 1 = Minor/Mild Improvement (0.25%), 2 = Moderate Improvement (26-50%), 3 = Marked Improvement (51-75%), 4 = Very Significant Improvement (76-100%) for Skin Laxity, Skin Texture, and Overall Appearance for the upper face, middle face, lower face, and neck.

OTHER OUTCOMES:
Subject Global Aesthetic Improvement Scale | Month 6 post treatment
  The subject will make a direct visual assessment to grade the following indications using the below Quartile Improvement Scale: 0 = No improvement, 1 = Minor/Mild Improvement (0.25%), 2 = Moderate Improvement (26-50%), 3 = Marked Improvement (51-75%), 4 = Very Significant Improvement (76-100%) for Skin Laxity, Skin Texture, and Overall Appearance for the upper face, middle face, lower face, and neck.
Physician Global Aesthetic Improvement Scale | Month 6 post treatment
  The Investigator will make a direct visual assessment to grade the following indications using the below Quartile Improvement Scale: 0 = No improvement, 1 = Minor/Mild Improvement (0.25%), 2 = Moderate Improvement (26-50%), 3 = Marked Improvement (51-75%), 4 = Very Significant Improvement (76-100%) for Skin Laxity, Skin Texture, and Overall Appearance for the upper face, middle face, lower face, and neck.

CONTACTS AND LOCATIONS:
Overall Officials: Brian S Biesman, MD, Principal Investigator — The Practice of Brian S. Biesman, MD

IPD SHARING:
Plan to Share IPD: No